CLINICAL TRIAL: NCT02249052
Title: A Double Blind Study to Evaluate the Safety and Efficacy of Collagenase Clostridium Histolyticum (AA4500) in the Treatment of Lipoma
Brief Title: Double Blind Study to Evaluate the Efficacy of Collagenase Histolyticum in the Treatment of Lipoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerut, Zachary, M.D. (Individual)
Collaborators: Advance Biofactures Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-Lipoma II
Record Dates: First submitted 2014-08-18; First posted 2014-09-25 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-08

CONDITIONS: Lipoma
MeSH Terms: conditions — Lipoma | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 (Active Comparator): single injection of 0.58 mg study drug
  Interventions: Drug: AA4500
- Placebo (Placebo Comparator): single injection of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AA4500 — Subjects must present with 2 lipomas; one to receive AA4500 and one to receive placebo simultaneously
  Other Names: XIAFLEX, Collagenase Clostridium Histolyticum
  Arms: AA4500
Drug: placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether collagenase is effective in reducing the surface area of a subcutaneous benign lipoma.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of a Food and Drug Administration (FDA) approved drug (XIAFLEX) in the treatment of lipoma (fatty tumors). The fat in the lipoma is like normal fat except that it is enclosed in a balloon-like structure which is made of collagen (fibrous tissue). Treatment of the lipoma with an injection of XIAFLEX (a protein that breaks down collagen fibers) may dissolve the collagen/fibrous strands thereby decreasing the size of the lipoma or removing it. Each subject must have two lipomas; one lipoma to be treated with placebo and one lipoma to be treated with study drug, both to be observed similarly throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age, of either sex or any race
* Clinical history of at least 2 lipomas for at least one year
* Lipomas diagnosed as benign
* Two lipomas on distinctly separate parts of the body, or on the torso if 30 cm apart, with easily definable edges
* Each lipoma is a single mass with easily definable edges
* Lipomas are 5 to 24 cm squared
* Women of childbearing potential must use an acceptable method of birth control

Exclusion Criteria:

* Lipomas on the head, neck, hand or foot, or female breast
* Women who are nursing or pregnant
* Multi-lobular lipomas
* Subjects who have received an investigational drug within 30 days before receiving the first dose of study drug in this study
* Subjects with a known allergy to collagenase or any of the inactive ingredients in XIAFLEX
* Subjects with uncontrolled diabetes, hypertension, or thyroid disease, or any medical condition that would make the subject unsuitable for enrollment
* Subjects having prior treatment or trauma of the lipoma that could interfere with study assessments
* Subjects with a history of connective tissue diseases, rheumatological diseases
* Subjects taking anticoagulants or planning to receive anticoagulants (except for lo dose aspirin and over-the-counter nonsteroidal anti-inflammatory drugs) within 7 days of injection of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary E Gerut, MD, Principal Investigator — Private Practice
Locations (2):
- United States (2):
  - Aesthetic Center, Hewlett, New York
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at two study sites in the United States.
Pre-assignment Details: Subjects must present with 2 lipomas meeting inclusion criteria
Groups:
- AA4500 and Placebo: Each subject received a single injection of 1 mL containing 0.58 mg AA4500 in one lipoma and a single injection of 1 mL placebo in another lipoma
  Lipoma #1 was randomized to AA4500 or placebo with Lipoma #2 receiving the alternate intervention
Period: Overall Study
Arm/Group | AA4500 and Placebo
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AA4500 and Placebo: single injection of 0.58 mg study drug and placebo
  Subjects must present with 2 lipomas; one to receive AA4500 and one to receive placebo simultaneously
Arm/Group | AA4500 and Placebo
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (9.13)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Surface Area of the Lipoma at Six Months
Description: The primary efficacy outcome is lipoma visible surface area defined as the longest dimension ("length") times the longest dimension perpendicular to length ("width"). Visible surface area will be analyzed as the percent change from baseline at the 6-month visit.
Time Frame: Baseline and 6 months post injection
Population: All 19 subjects enrolled with 2 lipomas. All received AA4500 in one lipoma and placebo in the other lipoma.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- AA4500: Each subject received a single injection of 1 mL containing 0.58 mg AA4500
- Placebo: Each subject received a single injection of 1 mL placebo
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 19 | 19
percentage change from baseline | -81.277 (22.9) | 2.053 (12.1)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -83.330, 95% CI 2-sided [-95.394 to -71.265], Standard Deviation 25.0311

2. Secondary Outcome: Responder Analysis
Description: The number of participants with at least 50% decrease in visible lipoma surface area of lipoma relative to baseline
Time Frame: Baseline and 6 months
Population: All 19 participants
Measure: Number; unit: participants
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 19 | 19
participants | 17 | 0
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p < .0001, Sign test; Binomial proportion = .8947, 95% CI 2-sided [.6686 to .9870]

3. Secondary Outcome: Percent Change From Baseline in Greatest Dimension (Length) of Lipoma at 6 Months
Description: Change from baseline in lipoma length Calculated as the percent change from baseline for length of the lipoma treated with AA4500 and the lipoma treated with placebo.
Time Frame: Baseline and 6 months
Population: All study participants
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Groups:
- AA4500: Each participants received a single injection of 1 mL containing 0.58 mg AA4500
- Placebo: Each participant received a single injection of 1 mL placebo
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 19 | 19
Percent change from baseline | -64.1818 (28.97) | 0.156 (7.78)

4. Secondary Outcome: Subject Satisfaction
Description: Subjects very satisfied or somewhat satisfied with study treatment based upon Subject Questionnaire
Time Frame: 6 months
Population: 1 participant did not complete the questionnaire at the final visit; therefore the analysis population was based upon 18 participants
Measure: Number; unit: participants satisfied
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 18 | 18
participants satisfied | 18 | 7

5. Other Pre Specified Outcome: Change in Visible Surface Area
Description: Visible surface area is defined as the longest dimension ("length") times the longest dimension perpendicular to length ("width"). Visible surface area will be analyzed as the percent change from baseline.
Time Frame: 1 Month post injection
Population: All 19 subjects enrolled with 2 lipomas. All received AA4500 in one lipoma and placebo in the other lipoma.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 19 | 19
percentage change from baseline | -26.74 (35.57) | 0.174 (8.38)

6. Other Pre Specified Outcome: Change in Visible Surface Area
Description: as for outcome 5
Time Frame: 3 month post injection
Population: All 19 subjects enrolled with 2 lipomas. All received AA4500 in one lipoma and placebo in the other lipoma.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 19 | 19
percentage change from baseline | -62.51 (32.14) | 0.402 (12.92)

ADVERSE EVENTS:
Time Frame: 6 months post administration study medication
Description: Treatment emergent adverse events were collected after the date of administration of study medication through the last visit at 6 months post administration.
Arm/Group | AA4500 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=19) | Placebo (N=19)
Injection site Bruising (General disorders) | 17 (17) | 3 (3) — Administration site condition
Injection site swelling (General disorders) | 15 (15) | 0 (0) — Administration site condition
Injection site pain (General disorders) | 10 (10) | 0 (0) — Administration site condition
Injection site pruritis (General disorders) | 4 (4) | 0 (0) — Administration site condition
Injection site haemorrhage (General disorders) | 2 (2) | 0 (0) — Administration site condition
Injection site discolouration (General disorders) | 1 (1) | 0 (0) — Administration site condition
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.